CLINICAL TRIAL: NCT05616962
Title: Vasculera in Participants With Lipedema an Exploratory Controlled Case Study
Brief Title: Vasculera in Participants With Lipedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLP-01
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-06

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Intervention Model Description: three (3) month open-label case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vasculera (Other): Vasculera 630 milligrams, two times per day
  Interventions: Dietary Supplement: Diosmiplex

INTERVENTIONS:
Dietary Supplement: Diosmiplex — diosmin glycoside in combination with alkaline granules known as alka4-complex
  Other Names: Vasculera

SUMMARY:
This study is designed to gain preliminary information via a uniform protocol regarding the clinical effects of Vasculera in participants with lipedema and the possible role of the glycocalyx as a physiological target for Vasculera activity. It is anticipated that the results of this case study will inform the development of a formal randomized, double-blind, placebo controlled trial.

DETAILED DESCRIPTION:
The goal of this type of clinical trial is to compare the measurement of participants legs before treatment and after using the treatment for approximately 3 months in clinic patients 20 to 70 years old with lipedema. The main questions it aims to answer are: does the leg circumference decrease and does the participants' overall wellbeing improve?

Participants will:

* Have physical examinations and measurements at baseline and 3 month visit
* Complete wellbeing self-assessments at baseline and 3 month visit
* Have blood drawn for chemical markers at baseline and 3 month visit
* Complete four visits total

ELIGIBILITY:
Inclusion Criteria:

1. established diagnosis of lipedema for at least one (1) year
2. women, ages 20 to 70 years
3. score of at least 4 out of 10 on self-assessment on a 0-10 scale (10=worst) for overall sense of well being
4. be willing to stop compression therapy for one week prior to each visit

Exclusion Criteria:

1. other forms of leg enlargement, including lymphedema
2. any primary systemic vasculopathy
3. history of exposure to Vasculera or other diosmin containing medication within one (1) year of the screening visit
4. concomitant use of warfarin, platelet inhibitors, factor Xa inhibitors or any medication intended to reduce blood coagulability
5. concomitant use of diclofenac, metronidazole or chlorzoxazone
6. uncontrolled hypertension (BP>170/110), unstable cardiac disease, active skin ulceration
7. any other disease or condition that, in the opinion of the investigator, might put the
8. subject at risk by participation in this study OR confound evaluation of response to Vasculera
9. history of substance abuse within one (1) year of the screening visit or of current alcohol consumption more than one (1) unit daily. For purposes of this study, a unit of alcohol will be considered to be 12 oz of beer, 6 oz of wine or 1 oz of hard spirits.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, Study Director — Primus Pharmaceuticals
Locations (1):
- Primus Pharmaceuticals, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Article written by investigator Response to all queries
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 120 days from NCT assignment
Access Criteria: Access will be given when requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 2 private medical offices between May 2019 and June 20219. The first participant first visit was May 26, 2019.
Pre-assignment Details: Of 34 participants recruited from site medical records, 34 met inclusion criteria and progressed to open-label treatment.
Period: Overall Study
Arm/Group | Vasculera
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vasculera: Vasculera 630 milligrams, one tablet two times per day
  Diosmiplex: diosmin glycoside in combination with alkaline granules known as alka4-complex
Arm/Group | Vasculera
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants] — Age was calculated from birthdate to informed consent
  Participants
    <=18 years | 0
    Between 18 and 65 years | 31
    >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants] — participant interview
  Participants
    Female | 34
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 7
  Race: White | 27
Weight [Mean (Standard Deviation); unit: Kilograms] | 102.54 (22.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline
Description: Weight in kilograms on digital, calibrated bathroom scale
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Vasculera
Number analyzed (Participants) | 34
kilograms | 0.340 (0.468)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.473, ANCOVA; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

2. Secondary Outcome: Percentage Change Right Leg at 2 Inches
Description: Right leg circumference measured at 2 inches above the right lateral malleoli
Time Frame: Visit 4 (3 month)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Vasculera
Number analyzed (Participants) | 18
percentage of change | -0.79 (1.44)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.03199, paired t-test

3. Secondary Outcome: Change in BMI From Baseline
Description: BMI in kilograms per meter squared
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: kilograms per meter squared
Arm/Group | Vasculera
Number analyzed (Participants) | 34
kilograms per meter squared | 0.14 (0.17)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.408, ANCOVA; ANCOVA with baseline value as covariate

4. Secondary Outcome: Change in Short Western Ontario and McMaster Universities Osteoarthritis Index Total Score From Baseline
Description: Short Western Ontario and McMaster Universities Osteoarthritis Index total score results calculated by summing the response to individual questions with range from 0 - 96 where 0 is the best score and 96 is the worst
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -7.12 (0.94)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — Reported p-value was calculated, did not attempt to indicate threshold for statistical significance. Significance was evaluated at <0.05. P-values were reported to the thousandths place and those less than 0.001 were reported as "<0.001"; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

5. Secondary Outcome: Change in Right Leg Discomfort From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.53 (0.39)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

6. Secondary Outcome: Change in Left Leg Discomfort From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.62 (0.37)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

7. Secondary Outcome: Change in Right Leg Feeling of Swelling or Tightness From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.65 (0.41)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

8. Secondary Outcome: Change in Left Leg Feeling of Swelling or Tightness From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.56 (0.47)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

9. Secondary Outcome: Change in Right Leg Tenderness From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.77 (0.46)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

10. Secondary Outcome: Change in Left Leg Tenderness From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.71 (0.48)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

11. Secondary Outcome: Change in Right Leg Bruising From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -3.44 (0.49)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

12. Secondary Outcome: Change in Left Leg Bruising From Baseline
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -3.26 (0.48)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

13. Secondary Outcome: Change in Right Leg Redness
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -1.79 (0.422)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

14. Secondary Outcome: Change in Left Leg Redness
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever seen or felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -1.85 (0.41)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

15. Secondary Outcome: Change in Fatigue
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -3.06 (0.40)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

16. Secondary Outcome: Change in Ability to Perform Activities of Daily Living
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.88 (0.40)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

17. Secondary Outcome: Change in the Overall Sense of Wellbeing
Description: An integer scale from 0 - 10 where 0 equals none and 10 equals worst ever felt
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | -2.47 (0.44)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Repeated measures ANCOVA with baseline value as covariate including the changes from Baseline to months 1, 2, and 3

18. Secondary Outcome: Investigator Assessment of Response to Therapy
Description: Likert scale from 0 to 5 where 0 is no response and 5 is the best response
Time Frame: Visit 4 (3 months)
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vasculera
Number analyzed (Participants) | 34
score on a scale | 3.29 (0.22)

19. Secondary Outcome: Percentage Change Right Leg at 12 Inches
Description: Right leg circumference measured at 12 inches above the right lateral malleoli
Time Frame: Visit 4 (3 month)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Vasculera
Number analyzed (Participants) | 18
percentage of change | -2.13 (2.78)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.00463, paired t-test

20. Secondary Outcome: Percentage Change Left Leg at 2 Inches
Description: Left leg circumference measured at 2 inches above the left lateral malleoli
Time Frame: Visit 4 (3 month)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Vasculera
Number analyzed (Participants) | 18
percentage of change | 0.73 (2.48)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.23077, paired t-test

21. Secondary Outcome: Percentage Change Left Leg at 12 Inches
Description: Left leg circumference measured at 12 inches above the left lateral malleoli
Time Frame: Visit 4 (3 month)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Vasculera
Number analyzed (Participants) | 18
percentage of change | 1.92 (2.74)
Statistical Analysis 1: Comparison: Vasculera; Test type: Superiority; p = 0.00849, paired t-test

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Vasculera
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

LIMITATIONS AND CAVEATS:
For 16 participants, the Change from Baseline could not be calculated as the Baseline measurement was incorrectly measured at 2 centimeters and 12 centimeters above the lateral maleoli and not 2 inches and 12 inches above the lateral maleoli per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT05616962/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT05616962/SAP_001.pdf